CLINICAL TRIAL: NCT02074852
Title: Comparison of Immediate Versus Delayed Removal of Urinary Catheter Following Elective Cesarean Section
Status: Completed | Type: Observational
Sponsor: Akmal El-Mazny (Other)
Responsible Party: Sponsor-Investigator, Akmal El-Mazny, Ass.Prof. , MD, Cairo University
Organization: Cairo University (Other)
Other Study IDs: urinary catheter following CS
Record Dates: First submitted 2014-02-24; First posted 2014-02-28 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Urinary Catheter; Cesarean Section; Urinary Infection
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Immediate catheter removal: The catheter was removed immediately after the CS
  Interventions: Other: Foley urethral catheter
- Delayed catheter removal: The catheter was removed 12 hours postoperatively
  Interventions: Other: Foley urethral catheter

INTERVENTIONS:
Other: Foley urethral catheter

SUMMARY:
The objective this trial is to compare immediate and 12 hours postoperative removal of urinary catheter after elective cesarean section; and whether early removal is associated with lower risk of urinary infection compared with delayed catheter removal.

ELIGIBILITY:
Inclusion Criteria:

- Women admitted to the prenatal wards for primary or repeat elective cesarean section

Exclusion Criteria:

* urinary infection (assessed clinically and by midstream urinalysis),
* significant vaginal bleeding,
* severe pre-eclampsia or eclampsia and/or any other conditions requiring postoperative monitoring of urinary output, and
* contraindications for general anesthesia.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women admitted to the prenatal wards for primary or repeat elective cesarean section
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of cases with significant bacteriuria and urinary symptoms | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Faculty of Medicine, Cairo University, Cairo, Egypt